CLINICAL TRIAL: NCT06556225
Title: Isolated Maxillary Sinus Lesions in Sohag University Hospital
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Karam Ali Alameldin, Isolated maxillary sinus lesions in Sohag university hospital, Sohag University
Other Study IDs: Soh-Med-24-04-018MS
Record Dates: First submitted 2024-07-20; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Maxillary Sinus Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of the study:

Identify variants of maxillary sinus pathologies, its clinical presentations, radiological findings and surgical managements.

DETAILED DESCRIPTION:
Maxillary sinus diseases are common and numerous disorders that affect this anatomical area. As lesions are frequently allowed to grow to a significant size before becoming symptomatic, patients often present late, which can make management options more limited and difficult. Proper evaluation both clinically and with appropriate imaging allows accurate diagnosis, and lesions can often be successfully managed endoscopically

ELIGIBILITY:
Inclusion Criteria:

* Only patients with isolated maxillary sinus lesions , with varying degrees of sinus opacity who were indicated for surgery.

Exclusion Criteria:

* Patients who had pan sinuses lesions or those with significant involvement of the other paranasal sinuses than maxillary sinus were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with the isolated maxillary sinus lesions were subjected to
  1. Detailed history, general clinical examination & ENT examination, routine investigations, diagnostic nasal endoscopy.
  2. CT scan PNS
  3. The surgical approaches and intraoperative findings were recorded either endoscopicallay or combined approach .
  4. The pathological diagnoses were reviewed postoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Identify variants of maxillary sinus pathologies, its clinical presentations, radiological findings and surgical managements. | will be at Sohag University Hospital, a tertiary care academic center in Egypt, from 2023 to 2024
  All the collected data will be analyzed using the Statistical Package for Social Sciences (SPSS) (SPSS Inc., Chicago, IL, USA)v22.

CONTACTS AND LOCATIONS:
Overall Officials: arafat mahmoud, Study Chair — sohag universty
Locations (1):
- Sohag Universty, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No